CLINICAL TRIAL: NCT01262326
Title: Determination of the Effect of Extreme Dietary Carbohydrate Restriction on Hepatic Glucose Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Browning, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 012005-053
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

ARMS (2):
- Low Carbohydrate Diet (Experimental): Subjects are placed on a low carbohydrate diet where only 5% of energy intake is derived from dietary carbohydrate.
  Interventions: Other: Calorie and Carbohydrate Restriction
- Low Calorie Diet (Active Comparator): Subjects have there caloric intake reduced to 1200 or 1500 kcal/day (women and men respectively).
  Interventions: Other: Calorie and Carbohydrate Restriction

INTERVENTIONS:
Other: Calorie and Carbohydrate Restriction — Carbohydrate Restriction = <20 g/d of dietary carbohydrate intake Calorie Restriction = 1200 kcal/d for women and 1500 kcal/d for men

SUMMARY:
All subjects will be evaluated by the Research Nurse at the Clinical Translational Research Center (CTRC) Outpatient Clinic to obtain informed consent, a brief medical history, weight, body mass index, waist/hip circumference and vital signs. Additionally, blood will be drawn at this visit to screen for renal dysfunction (Chem 10), liver disease (liver function tests (LFT's)), thyroid dysfunction (TSH), diabetes mellitus (HbA1C), and chronic inflammatory states (erythrocyte sedimentation rate). Subjects recruited to the study will be placed on a low-carbohydrate diet (<20 g/d without caloric restriction) designed either to promote weight loss or maintain weight stability for fourteen days prior to the protocol or they will consume a typical "Western" diet designed either to promote weight loss (restricted by 1300 kcal/d in the final fourteen days) or maintain weight stability for twenty-one days. Subjects recruited to the study will be lean, overweight, or obese and also may carry a diagnosis of NAFLD. Target accrual for total enrollment for this project will be set to 80 subjects to accommodate attrition and screen failures. The details of the low-carbohydrate diet have been discussed in consultation with Linda Brinkley, nutrition staff of the CTRC. Subjects chosen to undergo carbohydrate-restriction will have a teaching session with a CTRC dietician. Subjects will then initiate dietary carbohydrate-restriction on their own and keep a daily dietary record for seven days. At the end of seven days, the dietary record will be analyzed. The CTRC will then prepare all meals for the final seven days of the diet in accordance with daily caloric intake calculated from the dietary record. Calorie-restricted participants will keep a dietary record for one week while eating a typical "Western" diet. The dietician will analyze this record and meals restricted by 1300 kcal/d will be prepared by the CTRC for the final fourteen days of the diet. Alternatively, some subjects eating a typical "Western" diet may consume prepared meals with a fixed content of carbohydrate, fat, and protein that is unrelated to their pre-study dietary intake. In this scenario, the dietary carbohydrate content may be varied between 30 and 60% to provide information on differences in hepatic metabolism under conditions of differing, but clinically sustainable, carbohydrate intake. All participants will be admitted to the CTRC the night prior to the study and begin an overnight fast after dinner. Between 18:00 and 09:00, subjects will receive two stable isotope tracers orally: [U-13C]propionate at 08:00 (three 400 mg doses given over 1 hour) and 70% 2H2O at 22:00, 02:00, and 06:00. During the study subjects will also be given 0.5% 2H2O ad libitum. Two 500 mg acetaminophen tablets will also be given at 08:00. Between 08:00 and 09:00 subjects will undergo measurement of their respiratory quotient (RQ) using the CTRC indirect calorimeter (Delta Trac II).. Subjects will then have an intravenous catheter placed and an infusion of tracer amounts of [3,4-13C2]glucose, [1,2-13C]β-hydroxybutyrate and [3,4-13C]acetoacetate will be initiated. At 1 ½ and 2 hours after initiation of the infusion, a 50 cc blood draw will be performed. Voided urine will be collected every hour after ingestion of acetaminophen until the protocol concludes. The subject will then be given a meal and discharged from the CTRC, marking the completion of the protocol. The collected blood and urine will be transported by the research coordinator to the Advanced Imaging Research Center lab for analysis by MRS. Another blood draw (approximately 10 cc) will be done in conjunction with the final MRI in order to measure changes in the lipid profile after the diet intervention. The visits in their entirety will be as follows:

1 screening visit: 20 minutes

1. dietician visit: 20 minutes
2. MRS visits: 45 minutes each

1 (optional) overnight visit: 20 hours

ELIGIBILITY:
Inclusion Criteria:

The study will compare sources of hepatic glucose in individuals age 18 to 65 years matched for age, body mass index (BMI), gender, and ethnicity. Enrollment numbers will be higher to accommodate attrition and matching. The genders will be equally represented in both cohorts. The ethnicity of the participants will be chosen to match the general population in the Dallas area. Spanish speaking subjects will be eligible for enrollment. No cultural or ethnic background will be systematically excluded. The present study will be restricted to subjects who are overweight (25>BMI<35). All subjects will have a normal nutritional status and minimal ethanol intake (< 10 g/d). Because activity level is known to alter hepatic metabolism, the subjects chosen will be those who do not participate in regular exercise above the amount of activity associated with daily living. Participation in concurrent studies will be determined on a case-by-case basis. Informed consent will be obtained from all participants.

The investigators will also enroll subjects diagnosed with NAFLD from Dr. Browning's clinical hepatology practice.

Based upon the need to study the effects of macronutrient manipulation under a variety of conditions, the targeted enrollment for this protocol will be open-ended. This will allow the present application to act as the basis for studying hepatic metabolism under a variety of conditions. The enrollment target is 80 subjects.

Exclusion Criteria:

In order to eliminate confounding variables, the participants chosen will have to be in stable health, on no medications known to alter hepatic glucose metabolism, on no weight loss diet or diet pills within the previous 6 months, and without baseline ketonuria. The present study will be restricted to subjects who are overweight (25>BMI<35). Subjects with a history of renal calculi, gout/hyperuricemia, renal insufficiency, will also be excluded from the study. Pregnant women, children, and institutionalized individuals will also be excluded. NAFLD subjects with metal in or on their body will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-01; Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

PRIMARY OUTCOMES:
Liver triglyceride content | 2 weeks

SECONDARY OUTCOMES:
Measures of hepatic and whole-body oxidation | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Browning, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Result] Browning JD, Weis B, Davis J, Satapati S, Merritt M, Malloy CR, Burgess SC. Alterations in hepatic glucose and energy metabolism as a result of calorie and carbohydrate restriction. Hepatology. 2008 Nov;48(5):1487-96. doi: 10.1002/hep.22504. PMID 18925642
- [Derived] Browning JD, Baker JA, Rogers T, Davis J, Satapati S, Burgess SC. Short-term weight loss and hepatic triglyceride reduction: evidence of a metabolic advantage with dietary carbohydrate restriction. Am J Clin Nutr. 2011 May;93(5):1048-52. doi: 10.3945/ajcn.110.007674. Epub 2011 Mar 2. PMID 21367948